CLINICAL TRIAL: NCT00677105
Title: An Open-Label Phase I Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of JNJ-26481585 in Subjects With Advanced Stage and/or Refractory Solid Malignancies and Lymphomas
Brief Title: A Safety and Dose-finding Study of JNJ-26481585 for Patients With Advanced Solid Malignancies and Lymphoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013924
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Lymphoma; Neoplasms
Keywords: Lymphoma; Neoplasms; Solid Tumors; Advanced Cancer
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — quisinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: JNJ-26481585

SUMMARY:
The purpose of this study is to assess the safety of the drug (JNJ-24681585 a drug in development for cancer) in patients with advanced or refractory solid malignancies or lymphoma on the maximum dose that can be tolerated by these patients. The absorption, breakdown and elimination of the drug will be studied and in some patients, the effect of the food on these processes will also be examined.

DETAILED DESCRIPTION:
JNJ-24681585 is a histone deacetylase (HDAC) inhibitor. It is a drug in development for treatment of cancer. In this study, the safety (the effect on the body) of the drug in patients with advanced or refractory solid malignancies or lymphoma will be studied. The maximum dose that can be tolerated by patients will be determined. The absorption, break down, and elimination of the drug will be studied and in some patients the effect of food on these processes will be examined. Antitumor activity of JNJ-26481585 will be evaluated.

JNJ-26481585 will be administered in a continuous regimen with 21-day treatment cycles. The dose of JNJ-26481585 will start low and will be increased during the study in groups of 2 to 6 patients. The dose each patient receives at study entry will not increase, but patients who receive drug at a later enrollment time may receive a higher dose. If a group of patients does not have severe side effects, the next group of patients will get a higher dose. The dose will increase until some patients have severe side effects. The dose will then be decreased to a dose level where severe side effects are observed in less than 1/3 of patients. Once a safe dose level has been determined an additional group of 12-24 patients will be treated.

The amount of JNJ-26481585 in the blood will be measured and the effect on the disease will be evaluated in all patients. In some patients, the effect of food on the absorption, break down, and elimination of the study drug will also be studied.

Patients will be screened for eligibility within 4 weeks before study treatment is given. The treatment will consist of 21-day treatment cycles in a continuous once daily dosing regimen. The duration of treatment will depend on adverse effects and whether there is benefit from the treatment. The design of a cycle may be adjusted during the course of the study to include days when there is no treatment (a pause) as guided by clinical observations. The dosing regimen may be adjusted to twice daily or three times daily intake as guided by information on how rapidly your body breaks down and eliminates the study drug. Patients will be informed if there are changes in the design of a cycle or the dosing regimen.

During the first treatment cycle, patients are required to stay in the hospital for 3 or 4 nights. In addition there are 8 or 9 daytime visits during Cycles 1 and 2 (combined) that may take up to 12 hours after the morning dose at 2 or 3 occasions and up to 4 hours after the morning dose at the other 6 occasions. From Cycle 3 onwards, there is only 1 daytime visit per treatment cycle, and these visits usually take up less time.

Throughout the study, especially during Cycles 1 and 2, patients will undergo frequent blood and urine tests, procedures to assess safety including heart function, and tests to assess the course of the patients illness. Two weeks after the last dose of the study drug, patients are required to return to the study site for follow-up assessments. JNJ-26481585 will be provided as capsules and will be taken by mouth once daily throughout treatment. The starting dose level will be 2 mg but the dose received by an individual patient will be determined at the time of enrollment. Modifications to the treatment schedule or dosing regimen may be explored during the course of this study. Patients can continue receiving treatment as long as there is benefit as evaluated by the study doctor and there are no unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid malignancy or lymphoma that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective
* Performance status (based on the Eastern Cooperative Oncology Group assessments) of <= 2
* Life expectancy > 3 months
* Adequate gastrointestinal absorption status
* Adequate liver, kidney and bone marrow function
* Adequate heart function (Left Ventricular Ejection Fraction >= 50%)

Exclusion Criteria:

* Known brain metastases
* Chemotherapy (in the case of nitrosoureas and mitomycin C within 6 weeks), radiotherapy, immunotherapy or treatment with an investigational agent within 4 weeks before study drug administration
* History of uncontrolled heart disease or uncontrolled arterial hypertension (protocol-defined)
* Patients taking medications known to have a risk of causing heart function abnormalities (i.e.
* QTc prolongation and Torsades de Pointes)
* Neuropathy (malfunction of the nerves) at baseline of Grade > = 2
* Positive serology for Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Determine the safety and the maximum tolerated dose of JNJ-26481585. Determine how JNJ-26481585 and its metabolite, JNJ-26395018, are absorbed, broken down and eliminated after oral administration

SECONDARY OUTCOMES:
Investigate the effect of food on the absorption, break down and elimination of JNJ-26481585 and its metabolite, JNJ-26395018. Monitor the antitumor activity of JNJ-26481585.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (6):
- United Kingdom (6):
  - Glasgow
  - Leeds
  - London
  - Manchester
  - Newcastel Upon Tyne
  - Sutton